CLINICAL TRIAL: NCT01007994
Title: Reduction of Nocturnal Hypertension in Pediatric Renal Transplant Recipients
Brief Title: Reduction of Night-time Blood Pressure in Pediatric Renal Transplant Recipients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Christine B Sethna, MD, Division Director, Pediatric Nephrology, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09-054
Record Dates: First submitted 2009-11-04; First posted 2009-11-05 (Estimated); Results first posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Hypertension Secondary to Kidney Transplant
Keywords: Nocturnal hypertension; Pediatric; Renal Transplant; Pulse Wave Velocity; Echocardiogram; Pediatric Renal Transplant Recipient
MeSH Terms: interventions — Isradipine; Propranolol; Enalaprilat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- New Medication (Active Comparator): A new anti-hypertensive medication (enalapril, propranolol or isradipine) will be added at 8pm.
  Interventions: Drug: New Medication: Enalapril, Isradipine, Propranolol
- Control (No Intervention): Subjects in the control group will continue to take their medications as usual.

INTERVENTIONS:
Drug: New Medication: Enalapril, Isradipine, Propranolol — Enalapril will be added in the evening at 8 pm. If the subject is already on an ACEI or there is a contraindication to starting an ACEI the subject will be started on isradipine instead. If the subject is already on an ACEI and calcium channel blocker at baseline, propranolol will then be the new medication added.
  Dosing will be as follows:
  ACEI: Enalapril < 40 kg starting dose 2.5 mg titrate to 5 mg > 40 kg starting dose 5 mg titrate to 10mg Calcium Channel Blocker: Isradipine < 40 kg 2.5 mg > 40 kg starting dose 2.5 mg titrate to 5 mg Beta Blocker: Propranolol <40 kg starting dose 10 mg titrate to 20 mg >40 kg starting dose 20 mg titrate to 40 mg
  Other Names: Vasotec, DynaCirc, Inderal
  Arms: New Medication

SUMMARY:
The proposed study investigated the effect of chronotherapeutic alteration of anti-hypertensive medication on nocturnal hypertension and end-organ injury in pediatric renal transplant recipients who are non-dippers. Additionally, the investigators examined the association between response to intervention, serum adiponectin levels and adiponectin gene polymorphisms. The investigators hypothesized that (1) evening administration of anti-hypertensive medication will convert subjects from non-dipper to dipper status, improve mean nocturnal blood pressure (BP), and improve nocturnal BP load, (2) evening administration of anti-hypertensive medication will reduce albuminuria, left ventricular mass index (LVMI), rate of decline of glomerular filtration rate (eGFR) and will decrease pulse wave velocity (PWV).

DETAILED DESCRIPTION:
Study Design and Population A prospective, randomized, open label, blinded end-point (PROBE) pilot trial in pediatric kidney transplant recipients with non-dipping was conducted to determine the effect of chronotherapeutic alteration of anti-hypertensive medication on nocturnal BP. Non-dipper status was defined as <10% decline in systolic or diastolic BP from daytime to nighttime on ABPM. Participants were required to have a minimum of one follow-up study visit in order to be included in the analysis. Participants were recruited from Cohen Children's Medical Center in New Hyde Park, New York and from the Children's Hospital of Philadelphia (CHOP) in Philadelphia, Pennsylvania from 2010 to 2018.

Intervention Participants randomized to the treatment group were assigned to receive a new anti-hypertensive medication in the evening (1 hour prior to bed time) in addition to their regular baseline medications. The intervention medication was enalapril, an angiotensin converting enzyme inhibitor (ACEi). If the participant was already on an ACEi or there was a contraindication to starting an ACEi (e.g. hyperkalemia, history of allergic reaction to ACEi), then isradipine was added instead. If the participant was already on an ACEi and calcium channel blocker at baseline, then propranolol was the new medication added. The choice of medications was made based on the pharmacokinetic profile of the medications (quick-onset and short to intermediate acting) to lower nocturnal BP with evening administration. The dose of the new medication was titrated up to the target dose if the medication was tolerated and there were no adverse events reported at the two-week visit. Participants in the new medication group were evaluated at 2 weeks, 6 weeks, 3 months and 6 months by the study team to assess for side effects. Participants started on an ACEi had serum electrolytes, BUN and creatinine, and a pregnancy test monitored at each study visit. Participants with side effects were switched to a different class of medication. Participants randomized to the control group continued to take their medications as usual. Participants in the control group were followed at baseline, 3 months and 6 months. No changes to other BP medications were allowed during the 6-month study period. Any participant who developed hypertensive daytime casual BP on repeated measurements was withdrawn from the study.

Randomization and Blinding Participants were randomized in a 1:1 ratio to intervention or control arms in parallel utilizing a blocked randomization strategy (in blocks of 2 and 4) in order to ensure similar numbers of participants in each arm. The randomization scheme was computer generated. Group assignments were concealed in sealed envelops and randomization allocation was done sequentially by a person not directly involved with the study. Interpretation of the outcome data (ABPM, echocardiograms, PWV, labs) was adjudicated by investigators blinded to the treatment group. Laboratory technicians and echocardiographers were blinded to the participant treatment group.

Study Procedures Cardiovascular Measures 24-hour ABPM, echocardiography and PWV were performed at baseline, 3 months and 6 months. Echocardiography was performed using 2-D echo in M-mode in accordance with the recommendations of the American Society of Echocardiography. The SphygmoCor Vx PWV system (AtCor Medical Pty Ltd, Australia) was used to measure the velocity of the BP waveform between the carotid artery and the radial artery. Two PWV readings were obtained and the average was used for analysis. A 22-item pediatric sleep questionnaire was administered to the parent/guardian of the study subject to identify subjects with sleep-related breathing disorders. This questionnaire has been validated and tested for reliability in predicting obstructive sleep apnea. The Treatment Satisfaction Questionnaire for Medications (TSQM) was administered to assess patient satisfaction with the change in treatment and the impact of the therapy on quality of life. The tool gathers information about effectiveness of medication, side effects, convenience and global satisfaction, rated from 0-100 for each parameter.

Statistical Analysis Descriptive statistics were used to characterize demographic and clinical measures in participants. Fisher's exact test and Student's t-test were used to compare baseline variables between the treatment and control groups. Student's t-tests were used to compare continuous ABPM variables (nocturnal dip percent, mean BP, BP load) between treatment and control groups at 3 and 6 months post-intervention. Fisher's exact test was conducted to compare the proportion of participants who changed dipper status and nocturnal hypertension status between the two groups at 3 and 6 months. Within-person changes in each group were examined using the paired Student's t-test and McNemar's test. Student's t-test or Wilcoxon Rank Sum test for non-normally distributed variables were used to compare values of delta LVMI and eGFR between groups at each time point and paired tests for within-person changes. Intention-to-treat analysis was done. Statistical analyses was done using SPSS 25 (IBM Inc.) statistical package. A p-value < 0.05 was the criterion for statistical significance. For the primary outcome, the comparison of 14 subjects in each group provided 80% power (α = 0.05) to detect a 50% change from non-dipper status to dipper status in the treatment group compared to a 5% change in the control group. The study was not powered for analysis of secondary outcomes (LVMI, PWV, eGFR) as this was an exploratory aim for this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 5-21 years
* Stable kidney transplant recipients (<30% change in eGFR in past 3 months)
* eGFR > 30 ml/min/1.73 m2
* >6 months since kidney transplant
* ABPM: Non-dipper status defined as <10% decline in systolic or diastolic blood pressure from daytime to night-time

Exclusion Criteria:

* ABPM: Subjects with daytime mean blood pressure > 95% for height and sex
* Subjects on diuretic monotherapy will not be eligible for the time change group (to avoid discomfort of nocturnal enuresis)
* Subjects with nephrotic range proteinuria
* Subjects with major co-morbid conditions such as cardiac disease, pulmonary disease and diabetes mellitus
* Subjects/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures
* Subjects who are pregnant will not be eligible for the new medication group

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine B Sethna, MD, EdM, Principal Investigator — Northwell Health
Locations (2):
- United States (2):
  - Cohen Children's Medical Center of NY, New Hyde Park, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Natale P, Mooi PK, Palmer SC, Cross NB, Cooper TE, Webster AC, Masson P, Craig JC, Strippoli GF. Antihypertensive treatment for kidney transplant recipients. Cochrane Database Syst Rev. 2024 Jul 31;7(7):CD003598. doi: 10.1002/14651858.CD003598.pub3. PMID 39082471

RESULTS

PARTICIPANT FLOW:
Groups:
- New Medication: A new anti-hypertensive medication (enalapril, propranolol or isradipine) will be added at 8pm.
  New Medication: Enalapril, Isradipine, Propranolol: Enalapril will be added in the evening at 8 pm. If the subject is already on an ACEI or there is a contraindication to starting an ACEI the subject will be started on isradipine instead. If the subject is already on an ACEI and calcium channel blocker at baseline, propranolol will then be the new medication added.
  Dosing will be as follows:
  ACEI: Enalapril < 40 kg starting dose 2.5 mg titrate to 5 mg > 40 kg starting dose 5 mg titrate to 10mg Calcium Channel Blocker: Isradipine < 40 kg 2.5 mg > 40 kg starting dose 2.5 mg titrate to 5 mg Beta Blocker: Propranolol <40 kg starting dose 10 mg titrate to 20 mg >40 kg starting dose 20 mg titrate to 40 mg
Period: Overall Study
Arm/Group | New Medication | Control
Started | 17 | 16
Completed | 15 | 14
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | New Medication | Control | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.9 (4.3) | 14.3 (4.2) | 12.6 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 11 | 10 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 3 | 2 | 5
  Non-Black | 14 | 14 | 28
Left Ventricular Mass Index [Mean (Standard Deviation); unit: g/m^2.7] | 49.1 (14.1) | 39.7 (12.3) | 44.4 (13.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Are Non Dippers
Description: Percentage of subjects in each of the treatment arms who are nondippers, defined as systolic or diastolic nocturnal dip <10%
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | New Medication | Control
Number analyzed (Participants) | 17 | 16
Participants | 7 | 12

ADVERSE EVENTS:
Time Frame: 30 days after treatment duration of 6 months
Arm/Group | New Medication | Control
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 1/17 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | New Medication (N=17) | Control (N=16)
Hyperkalemia (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-25): https://cdn.clinicaltrials.gov/large-docs/94/NCT01007994/Prot_SAP_000.pdf